CLINICAL TRIAL: NCT02319148
Title: A Phase 1, Randomized, Open-label, 3-sequence, 4-treatment, Incomplete Block Design To Estimate The Effect Of Steady State Cyp3a4 Inhibitors (Itraconazole, Diltiazem Or Verapamil) On The Pharmacokinetics Of Singe Dose Pf-00489791 In Healthy Volunteers
Brief Title: A Study to Estimate the Effect of CYP3A4 Inhibitors (Itraconazole, Diltiazem or Verapamil) on the Pharmacokinetics of Single Dose PF- 00489791 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A7331022; 2014-001979-31 (EudraCT Number)
Record Dates: First submitted 2014-09-17; First posted 2014-12-18 (Estimated); Results first posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Itraconazole; Diltiazem; PF-00489791

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment B (Experimental): Treatment B subjects receive single dose administration of 20 mg PF-00489791 and multiple dose administration of itraconazole (200 mg once daily).
  Interventions: Drug: itraconazole; Drug: PF-00489791
- Treatment C (Experimental): Treatment C subjects receive single dose administration of 20 mg PF-00489791 and multiple dose administration of diltiazem (240 mg once daily).
  Interventions: Drug: diltiazem; Drug: PF-00489791
- Treatment D (Experimental): Treatment D subjects receive single dose administration of 20 mg PF-00489791 and multiple dose administration of verapamil (240 mg once daily).
  Interventions: Drug: SR verapamil; Drug: PF-00489791

INTERVENTIONS:
Drug: itraconazole — itraconazole dosed at 200 mg
  Arms: Treatment B
Drug: diltiazem — diltiazem dosed at 240 mg
  Arms: Treatment C
Drug: SR verapamil — SR verapamil dosed at 240 mg
  Arms: Treatment D
Drug: PF-00489791 — PF-00489791 20 mg single dose administration

SUMMARY:
The primary objective of the study is to estimate the effects of different strong enzyme (CYP3A4) inhibitors, itraconazole, diltiazem, or verapamil on the single dose pharmacokinetics of PF-00489791 in healthy volunteers. The study will enroll approximately 18 subjects that are randomized to 1 of 3 treatment groups. The study is also intended to determine the safety and tolerability of single-dose PF- 00489791 when it is administered with steady-state itraconazole, diltiazem, or verapamil.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests) with a Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs.) and with a personally signed and dated informed consent document and who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Participating female subjects of non-childbearing potential must meet at least one of the following criteria: achieved postmenopausal status; have undergone a documented hysterectomy and/or bilateral oophorectomy; have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations and females that do NOT have a documented hysterectomy, bilateral oophorectomy and/or ovarian failure) will be considered to be of childbearing potential.

Exclusion Criteria:

* Subjects cannot be included in the study if there is: the presence/ history of any disorder that prevents study completion
* Evidence/history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
* Any surgical or medical condition that may interfere with the absorption distribution, metabolism, or excretion of the study drug
* A positive urine drug screen or history of regular excessive alcohol consumption or use of tobacco-or nicotine-containing products in excess or from 24-hours prior to admission until discharge
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 halflives preceding the first dose of study med.
* Out of range blood pressure including current evidence of orthostatic change in blood pressure
* Abnormal ECG or history or current evidence of clinically important cardiac conduction abnormalities.
* Also excluded are: pregnant or breastfeeding female subjects; male subjects with partners currently pregnant; male and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as described in the protocol for the duration of the study and for at least 28 days after the last dose of investigational product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7331022&StudyName=A%20Study%20to%20Estimate%20the%20Effect%20of%20CYP3A4%20Inhibitors%20%28Itraconazole%2C%20Diltiazem%20or%20Verapamil%29%20on%20the%20Pharmacokinetics%20of%20Single%20Dose%20

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-00489791 20 mg: All participants who received a single-dose of PF-00489791 20 mg tablet orally during Period 1.
- PF-00489791 20 mg + Itraconazole 200 mg: All participants who received itraconazole 200 mg orally once daily for 7 days and a single-dose of PF-00489791 20 mg on Day 5 during Period 2.
- PF-00489791 20 mg + Diltiazem 240 mg: All participants who received diltiazem 240 mg MR tablet orally once daily for 13 days and a single-dose of PF-00489791 20mg on Day 11 during Period 2
- PF-00489791 20 mg + Verapamil 240 mg: All participants who received verapamil 240 mg SR tablet orally once daily for 13 days and a single-dose of PF-00489791 20 mg on Day 11 during Period 2.
Period: First Intervention Period
Arm/Group | PF-00489791 20 mg | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg
Started | 22 | 0 | 0 | 0
Completed | 22 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 4 Days
Arm/Group | PF-00489791 20 mg | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg
Started | 22 | 0 | 0 | 0
Completed | 22 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention Period
Arm/Group | PF-00489791 20 mg | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg
Started | 0 | 7 | 7 | 8
Completed | 0 | 6 | 6 | 6
Not Completed | 0 | 1 | 1 | 2
Not completed — Adverse event (AE) related to study drug | 0 | 0 | 1 | 1
Not completed — No longer willing to participate | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all eligible participants who received a single dose of PF-00489791 20 mg tablet orally.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg | Total
Number analyzed (Participants) | 7 | 7 | 8 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (6.1) | 33.4 (9.9) | 35.1 (10.1) | 35.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 7 | 7 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-00489791
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8 and 12 hours after PF-00489791 administration
Population: The pharmacokinetic (PK) analysis population included all participants randomized and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | PF-00489791 20 mg | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg
Number analyzed (Participants) | 22 | 6 | 6 | 6
nanograms per milliliter (ng/mL) | 1140 (34) | 1238 (33) | 1198 (33) | 1186 (21)
Statistical Analysis 1: Comparison: PF-00489791 20 mg vs PF-00489791 20 mg + Itraconazole 200 mg; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric means = 105.28, 90% CI 2-sided [92.11 to 120.34]
Statistical Analysis 2: Comparison: PF-00489791 20 mg vs PF-00489791 20 mg + Diltiazem 240 mg; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric means = 92.54, 90% CI 2-sided [80.96 to 105.77]
Statistical Analysis 3: Comparison: PF-00489791 20 mg vs PF-00489791 20 mg + Verapamil 240 mg; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric means = 116.36, 90% CI 2-sided [101.86 to 132.92]

2. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of PF-00489791
Description: AUC is a measure of the plasma concentration of the drug over time. It is used to characterize drug absorption.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8 and 12 hours after PF-00489791 administration
Population: The PK analysis population included all participants randomized and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-00489791 20 mg | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg
Number analyzed (Participants) | 22 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/mL) | 17880 (36) | 18140 (24) | 16840 (20) | 19560 (30)
Statistical Analysis 1: Comparison: PF-00489791 20 mg vs PF-00489791 20 mg + Itraconazole 200 mg; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric means = 90.16, 90% CI 2-sided [78.57 to 103.46]
Statistical Analysis 2: Comparison: PF-00489791 20 mg vs PF-00489791 20 mg + Diltiazem 240 mg; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric means = 106.38, 90% CI 2-sided [92.70 to 122.07]
Statistical Analysis 3: Comparison: PF-00489791 20 mg vs PF-00489791 20 mg + Verapamil 240 mg; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric means = 101.71, 90% CI 2-sided [88.68 to 116.66]

3. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-00489791
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8 and 12 hours after PF-00489791 administration
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hr/mL
Arm/Group | PF-00489791 20 mg | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg
Number analyzed (Participants) | 22 | 6 | 6 | 6
ng.hr/mL | 17580 (36) | 17980 (24) | 16760 (20) | 19400 (30)
Statistical Analysis 1: Comparison: PF-00489791 20 mg vs PF-00489791 20 mg + Itraconazole 200 mg; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric means = 91.33, 90% CI 2-sided [79.49 to 104.94]
Statistical Analysis 2: Comparison: PF-00489791 20 mg vs PF-00489791 20 mg + Diltiazem 240 mg; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric means = 106.97, 90% CI 2-sided [93.10 to 122.91]
Statistical Analysis 3: Comparison: PF-00489791 20 mg vs PF-00489791 20 mg + Verapamil 240 mg; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric means = 102.69, 90% CI 2-sided [89.42 to 117.93]

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-00489791
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8 and 12 hours after PF-00489791 administration
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | PF-00489791 20 mg | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg
Number analyzed (Participants) | 22 | 6 | 6 | 6
hour | 4.00 [2.00 to 4.08] | 3.50 [2.00 to 4.00] | 4.00 [1.00 to 4.00] | 4.00 [2.00 to 4.07]

5. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-00489791
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8 and 12 hours after PF-00489791 administration
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | PF-00489791 20 mg | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg
Number analyzed (Participants) | 22 | 6 | 6 | 6
liter | 18.06 (34) | 21.65 (18) | 19.98 (31) | 19.23 (23)

6. Secondary Outcome: Apparent Oral Clearance (CL/F) of PF-00489791
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8 and 12 hours after PF-00489791 administration
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per minute (mL/min)
Arm/Group | PF-00489791 20 mg | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg
Number analyzed (Participants) | 22 | 6 | 6 | 6
milliliter per minute (mL/min) | 18.64 (36) | 18.37 (24) | 19.81 (20) | 17.02 (30)

7. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of PF-00489791
Description: t1/2 is the time measured for the plasma concentration to decrease by one half.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8 and 12 hours after PF-00489791 administration
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-00489791 20 mg | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg
Number analyzed (Participants) | 22 | 6 | 6 | 6
hour | 11.39 (2.15) | 13.85 (2.79) | 11.75 (1.69) | 13.29 (2.56)

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities Meeting the Criteria for Potential Clinical Concern
Description: The following laboratory parameters were analyzed: hematology (hemoglobin, hematocrit, red blood cell [RBC] count, RBC morphology, platelet count, white blood cell [WBC] count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen [BUN], creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase [AST], alanine aminotransferase [ALT], total bilirubin, alkaline phosphatase, uric acid, albumin, and total protein; urinalysis (pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, microscopy [if urine dipstick was positive for blood, protein, nitrites or leukocyte esterase]); others (coagulation panel, circulating immune complex, and complement activation).
Time Frame: Baseline up to 28 days after last study drug administration
Population: The safety analysis population included all participants who received the study medication.
Measure: Number; unit: participants
Arm/Group | PF-00489791 20 mg | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg
Number analyzed (Participants) | 22 | 6 | 6 | 6
participants | 3 | 0 | 0 | 2

9. Secondary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Findings
Description: Vital signs assessment included pulse rate and blood pressure. Criteria for vital sign values meeting potential clinical concern included: supine/sitting pulse rate <40 or >120 beats per minute (bpm), standing pulse rate <40 or >140 bpm; systolic blood pressure (SBP) of >=30 millimeters of mercury (mm Hg) change from baseline in same posture or SBP <90 mm Hg, diastolic blood pressure (DBP) >=20 mmHg change from baseline in same posture or DBP <50 mm Hg.
Time Frame: Baseline up to Day 9
Population: The safety analysis population included all participants who received the study medication; n=number of participants evaluated against criteria.
Measure: Number; unit: participants
Arm/Group | PF-00489791 20 mg | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg
Number analyzed (Participants) | 22 | 7 | 7 | 8
participants
  Supine SBP <90 mm Hg (n=22,7,7,8) | 0 | 0 | 0 | 1
  Standing SBP <90 mm Hg (n=22,7,6,8) | 0 | 0 | 0 | 1
  Supine DBP <50 mm Hg (n=22,7,7,8) | 0 | 0 | 0 | 0
  Standing DBP <50 mm Hg (n=22,7,6,8) | 0 | 0 | 0 | 1
  Supine Pulse Rate <40 or >120 bpm (n=22,7,7,8) | 0 | 0 | 0 | 0
  Standing Pulse Rate <40 or >120 bpm (n=22,7,6,8) | 0 | 0 | 0 | 0
  Supine SBP >=30 mm Hg IFB (n=22,6,6,7) | 0 | 0 | 0 | 0
  Standing SBP >=30 mm Hg IFB (n=22,6,6,7) | 0 | 0 | 0 | 0
  Supine DBP >=20 mm Hg IFB (n=22,6,6,7) | 0 | 0 | 0 | 0
  Standing DBP >=20 mm Hg IFB (n=22,6,6,7) | 0 | 0 | 0 | 0
  Supine SBP >=30 mm Hg DFB (n=22,6,6,7) | 0 | 0 | 0 | 0
  Standing SBP >=30 mm Hg DFB (n=22,6,6,7) | 0 | 0 | 1 | 1
  Supine DBP >=20 mm Hg DFB (n=22,6,6,7) | 0 | 0 | 0 | 0
  Standing DBP >=20 mm Hg DFB (n=22,6,6,7) | 1 | 0 | 1 | 1

10. Secondary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Findings
Description: ECG parameters included PR interval, QRS interval, and corrected QT interval using Fridericia's formula (QTcF). Criteria for ECG changes meeting potential clinical concern included: PR interval greater than or equal to (>=)300 milliseconds (msec) or >=25% increase when baseline is greater than (>)200 msec and >=50% increase when baseline is less than or equal to (≤)200 msec; QRS interval >=140 msec or >=50% increase from baseline (IFB); and QTcF >=450 msec or >=30 msec increase. The number of participants with potentially clinically significant ECG findings at any visit were reported.
Time Frame: Pre-dose (Periods 1 and 2), 4, 72 and 96 hours post-dose in Period 2
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | PF-00489791 20 mg | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg
Number analyzed (Participants) | 22 | 7 | 7 | 8
participants
  PR Interval >=300 msec (n=22,7,7,8) | 0 | 0 | 0 | 0
  QRS Complex >=140 msec (n=22,7,7,8) | 0 | 0 | 0 | 0
  QTcF Interval 450-<480 msec (n=22,7,7,8) | 0 | 0 | 0 | 0
  QTcF Interval 480-<500 msec (n=22,7,7,8) | 0 | 0 | 0 | 0
  QTcF Interval >=500 msec (n=22,7,7,8) | 0 | 0 | 0 | 0
  PR Interval >=25/50% IFB (n=22,6,6,7) | 0 | 0 | 0 | 0
  QRS Interval >=50% IFB (n=22,6,6,7) | 0 | 0 | 0 | 0
  QTcF Interval 30-<60 msec IFB (n=22,6,6,7) | 0 | 1 | 0 | 0
  QTcF Interval >=60 msec IFB (n=22,6,6,7) | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants Who Used at Least 1 Concomitant Medication
Description: Participants were to abstain from all concomitant treatments, except for the treatment of AEs. Treatments taken after the first dose of study treatment were documented as concomitant treatments.
Time Frame: Baseline up to Day 15 (final study evaluation)
Population: The safety analysis population included all participants who received the study medication.
Measure: Number; unit: participants
Arm/Group | PF-00489791 20 mg | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg
Number analyzed (Participants) | 22 | 6 | 6 | 6
participants
  Drug Treatments | 10 | 2 | 4 | 2
  Non-Drug Treatments | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to 28 days after last study drug administration
Population: The safety analysis population included all participants who received the study medication.
Measure: Number; unit: participants
Groups:
- Itraconazole 200 mg: All participants who received itraconazole 200 mg orally once daily for 7 days.
- Diltiazem 240 mg: All participants who received diltiazem 240 mg MR tablet orally once daily for 13 days.
- Verapamil 240 mg: All participants who received verapamil 240 mg SR tablet orally once daily for 13 days.
Arm/Group | PF-00489791 20 mg | Itraconazole 200 mg | Diltiazem 240 mg | Verapamil 240 mg | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg
Number analyzed (Participants) | 22 | 7 | 7 | 8 | 6 | 6 | 6
participants
  AEs | 18 | 6 | 4 | 3 | 6 | 4 | 5
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last study drug administration
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-00489791 20 mg | Itraconazole 200 mg | Diltiazem 240 mg | Verapamil 240 mg | PF-00489791 20 mg + Itraconazole 200 mg | PF-00489791 20 mg + Diltiazem 240 mg | PF-00489791 20 mg + Verapamil 240 mg
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/7 | 0/7 | 0/8 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 18/22 | 6/7 | 4/7 | 3/8 | 6/6 | 4/6 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-00489791 20 mg (N=22) | Itraconazole 200 mg (N=7) | Diltiazem 240 mg (N=7) | Verapamil 240 mg (N=8) | PF-00489791 20 mg + Itraconazole 200 mg (N=6) | PF-00489791 20 mg + Diltiazem 240 mg (N=6) | PF-00489791 20 mg + Verapamil 240 mg (N=6)
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 4 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 14 | 1 | 4 | 2 | 6 | 4 | 2
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Spontaneous penile erection (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hot flush (Vascular disorders) | 3 | 0 | 0 | 0 | 5 | 2 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 1 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.